CLINICAL TRIAL: NCT04732273
Title: The Swiss Childhood Cancer Survivor Study - Follow-up (SCCSS-FollowUp)
Acronym: SCCSS-FU
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00739
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Late Effect; Childhood Cancer
Keywords: Childhood Cancer; Late Effects; Survivor
MeSH Terms: conditions — Neoplasms | interventions — Restraint, Physical; Health Records, Personal; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical examination, diagnostic tests, laboratory tests — Physical examination, diagnostic tests depending on examined organ system (e.g. lung function test, echocardiography, audiometry), and laboratory tests (e.g. kidney parameter, hormonal levels).
Other: Personal history, questionnaire — Personal history and focused questionnaires per organ system including symptoms, medication use, physical activity, and general wellbeing.

SUMMARY:
The SCCSS-FollowUp is a national, multicenter cohort study designed to investigate late effects in childhood cancer survivors in a prospective and longitudinal way. The study is embedded in regular follow-up care and inclusion in the study takes place in a step-wise approach. The investigators collect data from clinical examinations, laboratory and functional tests, and questionnaires to learn more about late effects of childhood cancer treatments.

DETAILED DESCRIPTION:
Background: Survival after childhood cancer has increased substantially over the last decades. In Switzerland, 10-year survival now exceeds 85%. This results in increasing numbers of childhood cancer survivors - estimated 6,600 survivors currently in Switzerland. Due to the cancer treatment or the cancer itself, a large part of the childhood cancer survivors suffer from late effects. As survivors of childhood cancer have decades of life ahead, it is of special interest to minimize potentially avoidable chronic diseases, impaired quality of life, deaths, and health care costs. There is a need to assess clinical data prospectively in a standardized way across clinics to study late effects on a national level. Such data are currently not available in Switzerland and the SCCSS-FollowUp aims to fill this gap.

Objectives: The SCCSS-FollowUp assesses the prevalence of late effects through risk-adapted medical examinations (in accordance with international guidelines and evidence), identifies CCS with asymptomatic late effects through functional testing, e.g. echocardiography or lung function testing, standardizes clinical follow-up examinations in CCS in Switzerland, and collects follow-up data in a longitudinal way. The SCCSS-FollowUp also investigates sociodemographic, treatment, lifestyle, and clinical risk factors for late effect development.

Methods: The SCCSS-FollowUp recruits eligible childhood cancer survivors in a stepwise approach by identifying CCS at risk because of specific treatment modalities (e.g. exposure to anthracyclines or thoracic irradiation). The investigators ask eligible survivors for participation. Those who consent receive before or during the next follow-up visits focused questionnaires. The questionnaires are short and focus on one organ system, but participants can receive different questionnaires at subsequent visits. The data generated during the follow-up visits, such as clinical examination, functional and laboratory test results, and the completed questionnaires are entered in the SCCSS-FollowUp database. The examinations and tests are performed in a standardized way in all participating clinics and according to follow-up guidelines or other evidence-based literature.

Rationale and significance:

The data collected within the SCCSS-FollowUp allow research on late effects on a national level and based on objective clinical data obtained during routine care. The SCCSS-FollowUp helps to learn more about late effects, especially subclinical damage, which are not detectable by questionnaire only. Early detection of these late effects and timely treatment can prevent and mitigate further deterioration. Furthermore, the SCCSS-FollowUp helps to assess risk factors for late effects development which can be used to amend cancer treatment in future patients. The SCCSS-FollowUp thus helps to improve the health of current and future childhood cancer survivors.

ELIGIBILITY:
This prospective cohort study is based on the Childhood Cancer Registry (ChCR), a national, population-based cancer registry that includes all children and adolescents in Switzerland who were diagnosed with cancer at age 0-20 years. It includes patients diagnosed with leukemia, lymphoma, central nervous system tumors, and malignant solid tumors or Langerhans cell histiocytosis.

Inclusion Criteria:

* Registered in the Childhood Cancer Registry (ChCR) or treated and followed-up in a Swiss pediatric oncology (SPOG) clinic, but not registered in the ChCR because of residency in neighboring countries
* Diagnosed at age 0 - 20 years
* Childhood cancer treatment completed
* All age categories at time of inclusion in the study (children, adolescents, adults)
* Written informed consent

Exclusion criteria:

* Childhood cancer survivors in a palliative or relapsed situation where no follow-up examinations are foreseen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Childhood cancer survivors, who were diagnosed in a Swiss pediatric oncology clinic at age <21 years from 1976 onward and who completed their cancer treatment. Survivors are eligible to participate to the study from the first day after treatment completion, but can also enter the study later.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2071-01-01 (Estimated); Study Completion 2071-01-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms of organ-specific late effects (example of pulmonary late effects) | At baseline
  Number of people with cough or shortness of breath when at risk for pulmonary late effects
Signs of organ-specific late effects (example of pulmonary late effects) | At baseline
  Number of people with signs of disturbed breathing or abnormal breathing sounds when at risk for pulmonary late effects
Tests to assess organ-specific late effects (example of pulmonary late effects) | At baseline
  Number of people with abnormal pulmonary function testing (e.g. spirometry, body plethysmography) when at risk for pulmonary late effects

SECONDARY OUTCOMES:
Symptoms of organ-specific late effects (example of pulmonary late effects) | 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Number of people with cough or shortness of breath when at risk for pulmonary late effects
Signs of organ-specific late effects (example of pulmonary late effects) | 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Number of people with signs of disturbed breathing or abnormal breathing sounds when at risk for pulmonary late effects
Tests to assess organ-specific late effects (example of pulmonary late effects) | 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Number of people with abnormal pulmonary function testing (e.g. spirometry, body plethysmography) when at risk for pulmonary late effects
Treatment-related risk factors for late effects | At baseline
  Cumulative dose of chemotherapeutic agents or radiotherapy, exposure to surgery and hematopoietic stem cell transplantation for each participant (not exhaustive)
Sociodemographic and socioeconomic characteristics potentially associated with late effects | At baseline, 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Collection of information on age at diagnosis, time since diagnosis, and gender for each participant (not exhaustive)
Lifestyle factors potentially associated with late effects | At baseline, 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Collection of information on smoking status, physical activity, and body mass index for each participant (not exhaustive)
Comorbidities potentially associated with late effects | At baseline, 1 year after recruitment, 2 years after recruitment, 3 years after recruitment, 4 years after recruitment, 5 years after recruitment, 10 years after recruitment, 15 years after recruitment, 20 years after recruitment
  Collection of information on arterial hypertension or obesity for each participant (not exhaustive)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, MD, Principal Investigator — Institute of Social and Preventive Medicine, University of Bern
Locations (3):
- Switzerland (3):
  - University Childen's Hospital Basel, Basel
  - University Children's Hospital Bern, Bern
  - University Hospital Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarkovic M, Schindera C, Sommer G, Schneider C, Usemann J, Otth M, Luer S, Ansari M, Latzin P, Kuehni CE. Assessing Pulmonary Function in Children and Adolescents After Cancer Treatment: Protocol for a Multicenter Cohort Study (Swiss Childhood Cancer Survivor Study FollowUp-Pulmo). JMIR Res Protoc. 2025 Apr 8;14:e69743. doi: 10.2196/69743. PMID 40198919